CLINICAL TRIAL: NCT05990803
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 Monotherapy, SI-B003 Monotherapy and BL-B01D1+SI-B003 Combination Therapy (BL-B01D1+SI-B003) in Patients With Recurrent or Metastatic Cervical Cancer and Other Gynecological Malignancies
Brief Title: A Study of BL-B01D1, SI-B003 and BL-B01D1+SI-B003 in Patients With Recurrent or Metastatic Cervical Cancer and Other Gynecological Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-SI-B003-201-08
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer
Keywords: Gynecological malignancies
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants received BL-B01D1, SI-B003 or BL-B01D1 + SI-B003 therapy in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-B01D1; Drug: SI-B003

INTERVENTIONS:
Drug: BL-B01D1 — BL-B01D1 was administered by intravenous infusion on D1 and D8 in a 3-week cycle.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: SI-B003 — SI-B003 was administered by intravenous infusion every 3 weeks (Q3W).

SUMMARY:
Objective: To explore the efficacy, safety and tolerability of BL-B01D1, SI-B003 and BL-B01D1+SI-B003 in patients with recurrent or metastatic cervical cancer and other gynecological malignancies, and to further explore the optimal dose and mode of combination.

DETAILED DESCRIPTION:
Objective: To explore the efficacy of BL-B01D1 monotherapy, SI-B003 monotherapy, and BL-B01D1+SI-B003 combination therapy in patients with recurrent or metastatic cervical cancer. To explore the safety and tolerability of BL-B01D1 monotherapy, SI-B003 monotherapy and BL-B01D1+SI-B003 combination therapy in patients with recurrent or metastatic cervical cancer and other gynecological malignancies, and to further explore the optimal dose and mode of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject volunteered to participate in the study and signed an informed consent;
2. Women aged ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG score 0-1;
5. Gynecological malignancies such as recurrent or metastatic cervical cancer confirmed by histopathology and/or cytology after failure or intolerance to standard treatment or for which no standard treatment is available;
6. Agree to provide 10 surgical specimens or fresh tissue samples of primary or metastatic tumors within 3 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. No blood transfusion, colony-stimulating factor, any cell growth factor injection, or albumin injection were allowed within 14 days before the first use of the study drug, and the organ function level must meet the requirements;
9. Urine protein ≤2+ or ≤1000g/24h;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
12. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, a serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Prior treatment with an ADC drug with a topoisomerase I inhibitor as a toxin;
2. Use of antineoplastic therapy within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral fluorouracil or palliative radiotherapy within 2 weeks before the first dose;
3. Cohort_B and Cohort_C with a history of immunotherapy and grade ≥3 irAE or grade ≥2 immune-related myocarditis;
4. Cohort_B, Cohort_C, who had received an immunomodulatory drug within 14 days before the first dose of study drug;
5. Had a history of serious cardiovascular and cerebrovascular diseases;
6. Active autoimmune and inflammatory diseases;
7. Other malignant tumors that progressed or required treatment within 5 years before the first dose;
8. A history of ILD requiring steroid therapy, current ILD, or suspected ILD at screening that could not be ruled out by imaging;
9. History of poorly controlled diabetes mellitus, poorly controlled hypertension, or hypertensive crisis or hypertensive encephalopathy before the first medication;
10. New onset of deep vein thrombosis within 14 days before screening or pulmonary embolism within 6 months;
11. Patients with active central nervous system metastases;
12. Patients with massive, symptomatic, poorly controlled, or unstable effusions;
13. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any of BL-B01D1's excipients;
14. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation;
15. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
16. Active infections requiring systemic therapy, such as severe pneumonia, bacteremia, sepsis, etc;
17. Had participated in another clinical trial within 4 weeks before the first dose;
18. Who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
19. Patients with a history of intestinal obstruction within 6 months before the screening period;
20. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study .

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, PHD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China